CLINICAL TRIAL: NCT02044679
Title: Evaluation of Spot Urine as a Biomarker of Fluid Intake in Real Life Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NU365
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A = Increase water intake 1 (Experimental): + 1,5 to 2,0 L/day of water
  Interventions: Other: Water
- B = Increase water intake 2 (Experimental): + 1,0 to 1,5 L/day of water
  Interventions: Other: Water
- C = no change (Other): No change
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Water
  Arms: A = Increase water intake 1; B = Increase water intake 2
Other: No intervention
  Arms: C = no change

SUMMARY:
Evaluate urine osmolality as a marker of fluid intake, in healthy subjects displaying a wide range of fluid intake behaviors

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male subjects aged 20- 30 years old (both ages included).
* BMI within the range 20-25 kg/m2 (both inclusive).
* Height within the range 1.60-1.75 m (both inclusive) for female subjects and 1.70-1.85 m (both inclusive) for male subjects.
* Monophasic contraceptive method (female subjects only)
* Smoking less than 10 cigarettes/day
* Fluid intake habits falling within one of three designated arms

Exclusion Criteria:

* Pregnant woman (as determined by a pregnancy test) or woman planning to become pregnant during the study; breast-feeding woman.
* Any clinically relevant acute or chronic diseases which could interfere with the subjects' safety during the trial, or expose them to undue risk, or which could interfere with the study objectives.
* Having participated in a clinical study for the renal diseases or having received any treatment related to the kidneys, cardiovascular disease or to hypertension in the last 12 months.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Osmolality | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- BIOTRIAL, Rennes, France

REFERENCES:
- [Derived] Lemetais G, Melander O, Vecchio M, Bottin JH, Enhorning S, Perrier ET. Effect of increased water intake on plasma copeptin in healthy adults. Eur J Nutr. 2018 Aug;57(5):1883-1890. doi: 10.1007/s00394-017-1471-6. Epub 2017 Jun 3. PMID 28578535